CLINICAL TRIAL: NCT01674816
Title: (Étude de la cinématique Tridimensionnelle du Genou et Guidage Chirurgical Minimalement Effractifs Par Recalage Rigide échographique)
Brief Title: Minimally Invasive Three-dimensional Knee Kinematic Assessment and Surgical Guidance Using Ultrasonic Rigid Registration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Eiffel Medtech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE12.006
Record Dates: First submitted 2012-08-06; First posted 2012-08-29 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis; Knee Instability; 3D Knee Kinematics; Precision of Surgical Actions; Clinical Outcomes
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repeated Measurements of Knee Alignment and Kinematics (Active Comparator): Patients in the Repeated Measurements Arm will have the kinematic measurement protocol repeated twice before and twice after the surgical procedure; the procedure itself will be performed with the traditional technique, i.e without guidance by the system.
  Interventions: Device: Repeated Measurements of Knee Alignment and Kinematics
- Computer Guidance of Surgical Actions (Active Comparator): Patients in the Computer Guidance of Surgical Actions Arm will have the kinematic measurement protocol performed only once before and once after the surgical procedure; the procedure itself will be performed with guidance by the system.
  Interventions: Device: Computer Guidance of Surgical Actions

INTERVENTIONS:
Device: Repeated Measurements of Knee Alignment and Kinematics — Repeated Measurements of Knee Alignment and Kinematics using tools developed by Eiffel Medtech Inc.
  Arms: Repeated Measurements of Knee Alignment and Kinematics
Device: Computer Guidance of Surgical Actions — Computer Guidance of Surgical Actions using tools developed by Eiffel Medtech Inc.
  Arms: Computer Guidance of Surgical Actions

SUMMARY:
Problem:

Currently, no system allows precise kinematic assessment of the knee and accurate guiding of orthopedic surgical actions in a minimally invasive fashion. However, such a system would prove useful in the clinical setting to improve the quality of surgical interventions at the knee.

Hypothesis:

A novel knee kinematic assessment and surgical guidance tool using 3D personalized imaging and minimally invasive bony fixation allows precise kinematic assessment and surgical guidance in the routine clinical setting.

Objectives :

* Demonstrating the capacity of the system to precisely measure 3D knee kinematics
* Quantifying the reproducibility of the kinematic measurements
* Measuring the impact of knee surgical procedures on knee kinematics
* Assessing the correlations between measured articular kinematics and clinical results after knee surgery
* Integrating the novel measuring system to the surgical flow of three knee surgical procedures
* Quantifying the precision and reproducibility of the surgical actions guided by the system
* Comparing the clinical results of surgeries guided by the system to those performed with the traditional technique

DETAILED DESCRIPTION:
A novel knee kinematic assessment and surgical guidance tool using 3D personalized imaging and minimally invasive bony fixation allows precise kinematic assessment and surgical guidance in the routine clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients awaiting a knee surgery (total knee arthroplasty (TKA), high tibial osteotomy (HTO), anterior cruciate ligament reconstruction(ACLR))

Exclusion Criteria:

* Active infection
* Atypical morphology and/or alignment of the lower limbs
* Knee instability (other than secondary to ACL deficiency in patients awaiting ACLR)
* Knee flexion contracture of 10 degrees or more
* Knee flexion of less than 120 degrees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
3D knee kinematic assessment | 1 day
  The system should be able to precisely and reproducibly measure 3D knee kinematics (tibio-femoral flexion, abduction-adduction, transverse rotation, and anterio-posterior and medio-lateral translations)
Precision of guided surgical actions | During surgery
  The system should allow the surgeon to realize surgical actions, like bone cuts and guide-wire placement, within one degree and one millimeter of the desired target.
Precision of guided surgical actions | On post-operative imaging (six weeks after surgery)
  The system should allow the surgeon to realize surgical actions, like bone cuts and guide-wire placement, within one degree and one millimeter of the desired target.

SECONDARY OUTCOMES:
Clinical results | At each post-operative visit (six weeks, six months, one year, and two years after surgery)
  The clinical results after surgery will be assessed using patient questionnaire and clinical examination.
Clinical results | At each post-operative visit (six weeks, six months, one year, and two years after surgery)
  The clinical results after surgery will be assessed using the International Knee Society score.
Clinical results | At each post-operative visit (six weeks, six months, one year, and two years after surgery)
  The clinical results after surgery will be assessed using the KOOS score.
Clinical results | At each post-operative visit (six weeks, six months, one year, and two years after surgery)
  The clinical results after surgery will be assessed using the SF-12 score.
Clinical results | At each post-operative visit (six weeks, six months, one year, and two years after surgery)
  The clinical results after surgery will be assessed using the Marx activity scale.
Clinical results | At each post-operative visit (six weeks, six months, one year, and two years after surgery)
  The clinical results after surgery will be assessed through angular and linear measurements using 3D imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lavoie, MD, MSc, FRCSC, Principal Investigator — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada